CLINICAL TRIAL: NCT00652184
Title: Phase 2/3 Multi-Center, Double-Blind, Controlled Trial Comparing Topical ARYS-01 (Sorivudine) Cream 3%, Oral Valaciclovir, and Combination Topical ARYS-01 Cream /Oral Valaciclovir for Treatment of Herpes Zoster in Immunocompetent Patients 18 Years of Age or Older
Brief Title: Study to Compare Efficacy of Topical ARYS-01 (Sorivudine) Cream 3%, Oral Valaciclovir and Combination ARYS-01 Cream 3%/Oral Valaciclovir for Treatment of Herpes Zoster (Shingles)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: aRigen Pharmaceuticals, Inc. (Industry)
Responsible Party: President and Chief Executive Officer, aRigen Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARYS-0701
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-10

CONDITIONS: Herpes Zoster; Postherpetic Neuralgia
Keywords: antiviral; herpes zoster; postherpetic neuralgia; varicella zoster virus; shingles
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic; Chickenpox | interventions — sorivudine; Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Placebo cream BID for 10 days and placebo valaciclovir caplets TID from days 1-3 and active valaciclovir caplets 1 gram TID from days 4-10
  Interventions: Drug: placebo; Drug: valaciclovir
- 2 (Active Comparator): Placebo cream BID for 10 days and active valaciclovir caplets TID from days 1-10
  Interventions: Drug: ARYS-01 (sorivudine) cream 3% or placebo cream; Drug: placebo; Drug: valaciclovir
- 3 (Experimental): Active cream BID for 10 days and placebo valaciclovir caplets TID from days 1-3 and active valaciclovir caplets 1 gram TID from days 4-10
  Interventions: Drug: ARYS-01 (sorivudine) cream 3% or placebo cream; Drug: placebo; Drug: valaciclovir
- 4 (Other): Active cream BID for 10 days and active valaciclovir caplets TID from days 1-10
  Interventions: Drug: ARYS-01 (sorivudine) cream 3% or placebo cream; Drug: valaciclovir

INTERVENTIONS:
Drug: ARYS-01 (sorivudine) cream 3% or placebo cream — sorivudine cream 3% or placebo cream twice daily for 10 days
  Other Names: ARYS-01 cream 3%; sorivudine cream 3%; topical sorivudine 3%
  Arms: 2; 3; 4
Drug: placebo — placebo cream and placebo valaciclovir
  Arms: 1; 2; 3
Drug: valaciclovir — active valaciclovir

SUMMARY:
A multi-center, randomized, 4-arm, placebo-controlled, double-blind efficacy study of ARYS-01 (sorivudine) cream 3%.

DETAILED DESCRIPTION:
More than 95% of people are infected with varicella Zoster virus (VZV) at one time of life or another. Primary VZV infection manifests as varicella (chicken pox). The virus then establishes a latent infection of the sensory ganglia from which it may reactivate years later to produce the clinical syndrome of Herpes Zoster (shingles). The initial cutaneous VZV lesions are pruritic, erythematous macules; and the lesions progress through maculopapular stage to vesicular, ulceration and crusting phases. The crusting phase signals the beginning of the healing process, and begins with clouding of the vesicular fluid, within about 24 to 48 h after the appearance of each lesion. This is a Phase 2 study to assess: 1) the overall benefit of ARYS-01 (sorivudine) cream 3% vs. Placebo cream (with immediate or delayed use of Valaciclovir therapy) on Herpes Zoster rash healing rates and postherpetic neuralgia (PHN), 2) the efficacy of ARYS-01 cream 3% vs. Placebo cream, prior to initiation of Valaciclovir, to build evidence for monotherapy treatment benefit of ARYS-01 cream on the initial onset of Herpes Zoster symptoms, 3) the efficacy of ARYS-01 cream 3% vs. Placebo cream, with immediate or delayed initiation of Valaciclovir, for synergetic effects on the initial onset of Herpes Zoster symptoms.

The primary efficacy endpoint is the effect of ARYS-01 cream (with or without Valaciclovir) on the reduction of the crusting stage of VZV rash present at Day 8. Secondary endpoints include time to cessation of new lesion formation, and time to cessation of Zoster-associated pains, pain intensity, rash healing and size reduction, and lesion dissemination.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* diagnosed with herpes zoster
* confirmed for VZV with lesion swab at screening and subsequent PCR test.
* contraception for women of child-bearing potential
* be able to communicate with investigator and compliant

Exclusion Criteria:

* cytotoxic or immunosuppressive drugs within 3 mos, 5-FU or its pro-drugs, tricyclic antidepressants, probenecid, topical or systemic antiviral drugs or immunomodulatory agents for viral infection
* herpes zoster ophthalmicus
* female patients who are pregnant and/or nursing or planning a pregnancy
* congenital, acquired or corticosteroid-induced immunodeficiency, including malignancy
* renal insufficiency or creatinine level >2mg/dL
* clinical significant liver enzyme abnormalities and any other laboratory abnormalities determined by the screening lab
* history of intolerance or hypersensitivity to the cream components
* current significant skin disease within affected dermatome
* history of positive result for hepatitis B surface antigen, hepatitis C virus, or HIV
* current participation in another clinical drug research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-06 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
The effect of ARYS-01 (sorivudine) cream (with or without Valaciclovir) on the reduction of the crusting stage of VZV rash present at Day 8. | Day 8

SECONDARY OUTCOMES:
The time to cessation of new lesion formation, and time to cessation of Zoster-associated pains, pain intensity, rash healing and size reduction, and lesion dissemination. | Day 4

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - ARYS-0701 Site 3, Beverly Hills, California
  - ARYS-0701 Site 6, Encino, California
  - ARYS-0701 Site 7, Vista, California
  - ARYS-0701 Site 8, Henderson, Nevada
  - ARYS-0701 Site 9, Las Vegas, Nevada
  - ARYS-0701 Site 10, New York, New York
  - ARYS-0701 Site 11, New York, New York
  - ARYS-0701 Site 4, New York, New York
  - ARYS-0701 Site 12, Raleigh, North Carolina
  - ARYS-0701 Site 1, Houston, Texas

REFERENCES:
- [Derived] Satyaprakash AK, Tremaine AM, Stelter AA, Creed R, Ravanfar P, Mendoza N, Mehta SK, Rady PL, Pierson DL, Tyring SK. Viremia in acute herpes zoster. J Infect Dis. 2009 Jul 1;200(1):26-32. doi: 10.1086/599381. PMID 19469706